CLINICAL TRIAL: NCT04481997
Title: Anti-thrombotic and Glucose loweRing THerapy in diabEtics With CAD Undergoing PCI: a Prospective Multicenter observatIonal Study on Their Use and Implications for Clinical Outcomes - The ARTHEMIS Registry
Brief Title: Anti-thrombotic and Glucose Lowering Therapy in Diabetic Patients Undergoing PCI
Acronym: ARTHEMIS
Status: Completed | Type: Observational
Sponsor: Associacao para Investigacao e Desenvolvimento da Faculdade de Medicina - CETERA (Other)
Collaborators: AstraZeneca (Industry); Cardiovascular Centre of Universidade de Lisboa (CCUL) (Unknown)
Responsible Party: Sponsor
Other Study IDs: CET.NIS2020.01; ESR-19-20188 (Other Grant/Funding Number: AstraZeneca)
Record Dates: First submitted 2020-06-26; First posted 2020-07-22 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Type2 Diabetes Mellitus; Coronary Heart Disease
Keywords: PCI-Percutaneous Coronary Intervention; Diabetes Mellitus; Dual Antiplatelet Therapy; Anti-diabetic drugs
MeSH Terms: conditions — Coronary Disease; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Diabetic patients with CAD submitted to PCI: Individuals with type 2 Diabetes mellitus (previously diagnosed or diagnosed at index admission) submitted to PCI
  Interventions: Other: Exposure to Anti-thrombotic treatment agents and glucose lowering therapy

INTERVENTIONS:
Other: Exposure to Anti-thrombotic treatment agents and glucose lowering therapy — Exposure to Anti-thrombotic treatment agents and glucose lowering therapy

SUMMARY:
Diabetes mellitus (DM) is one of the main risk factors for ischemic events in patients with coronary artery disease (CAD) and diabetes is a factor in several post-PCI (Percutaneous Coronary Intervention) risk scores. However, until recently, there were almost no studies performed specifically in the diabetic population of patients undergoing PCI. This study aims to describe the anti-thrombotic regimens, clinical outcomes and current diabetes medical treatment in an unselected consecutive population of patients with DM undergoing PCI.

DETAILED DESCRIPTION:
Diabetes is one of the main risk factors for ischemic events in patients with coronary artery disease and diabetes is a factor in several post-PCI risk scores (including the commonly used DAPT score). However, until recently, there were almost no studies performed specifically in the diabetic population of patients undergoing PCI. At large, results from randomized trials assessing the duration of DAPT have produced conflicting results and there is uncertainty about the best anti-thrombotic strategy in patients with diabetes. Further assessment of the patterns of use and their clinical effects, including those related to prolonged DAPT is needed, in diabetic patients, especially in less selected "real world" populations.

ELIGIBILITY:
Inclusion Criteria:

* PCI with stent implantation, performed in at least one major coronary artery in the context of stable coronary artery disease or acute coronary syndrome
* Type 2 Diabetes mellitus (previously diagnosed or diagnosed at the index admission)
* Informed consent signed
* Patient not simultaneously participating in any interventional study

Exclusion Criteria:

* Patients with Type 1 Diabetes mellitus
* Patients whose survival is expected to be lower than 1 year at hospital discharge
* Patients not whiling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1000 Type 2 Diabetes mellitus consecutive patients submitted to PCI in 12 interventional Cardiology Portuguese centers
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2023-11-04 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Enumeration of the anti-thrombotic agents prescribed to patients | Baseline to 24 months follow-up
Planned duration of dual anti-platelet treatment (DAPT) after the PCI. | From index admission to 24 months follow-up
Adherence to anti-thrombotic regimen | 6 to 24 months follow-up
  Classified qualitatively according to the assessment of the attending physician.
Actual duration of DAPT (if different from the planned duration) | 6 to 24 months follow-up
Reasons for interrupting DAPT at a time different from the planned duration | 6 to 24 months follow-up
Reasons for prolonging DAPT over 1 year | 12 to 24 months follow-up

SECONDARY OUTCOMES:
Major Adverse Coronary Events (MACE) | 6 to 24 months follow-up
  Major Adverse Coronary Events (MACE) (death from any cause, new spontaneous acute myocardial infarction, stroke).
Death rate from any cause | 6 to 24 months follow-up
Rate of cardiovascular death | 6 to 24 months follow-up
Rate of new spontaneous acute myocardial infarction | 6 to 24 months follow-up
Rate of hospital admissions for acute coronary infarction | 6 to 24 months follow-up
Rate of unplanned coronary revascularization | 6 to 24 months follow-up
Rate of stroke/transient ischemic attack | 6 to 24 months follow-up
Death rate from heart failure | 6 to 24 months follow-up
Rate of hospital admission due to heart failure | 6 to 24 months follow-up
Rate of bleeding events of type 3-5 of BARC (Bleeding Academic Research Consortium) scale | 6 to 24 months follow-up
  The BARC (Bleeding Academic Research Consortium) scale will be used. The minimum and maximum scores of the scale are, respectively, type 0 (no bleeding) and type 5 (fatal). There will only be collected the events corresponding to type 3-5 of BARC scale.
Rate of bleeding events of type 1-5 of BARC (Bleeding Academic Research Consortium) scale | 6 to 24 months follow-up
  The BARC (Bleeding Academic Research Consortium) scale will be used. The minimum and maximum scores of the scale are, respectively, type 0 (no bleeding) and type 5 (fatal). There will be collected the events corresponding to type 1-5 of BARC scale.
Percentage of patients treated with different glucose-lowering drugs. | Before index admission to 24 months follow-up.
Diabetes control (HbA1c values) | At baseline to 24 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Sérgio B Baptista, PhD, Principal Investigator — Cardiovascular Centre of the University of Lisbon (CCUL); Luís Raposo, MD, Principal Investigator — Hospital de Santa Cruz, CHLO, EPE, Lisbon, Portugal
Locations (12):
- Portugal (12):
  - Hospital de Braga, EPE, Braga, Braga District
  - Centro Hospitalar e Universitário de Coimbra - Hospital Geral & Hospital Universitário de Coimbra, Coimbra, Coimbra District
  - Centro Hospitalar Universitário do Algarve - Hospital de Faro, Faro, Faro District
  - Hospital Prof. Doutor Fernando Fonseca, Amadora, Lisbon District
  - Centro Hospitalar Lisboa Ocidental - Hospital de Santa Cruz, Carnaxide, Lisbon District
  - Centro Hospitalar Lisboa Central - Hospital de Santa Marta, Lisbon, Lisbon District
  - Centro Hospitalar Universitário Lisboa Norte - Hospital de Santa Maria, Lisbon, Lisbon District
  - Centro Hospitalar Universitário do Porto, EPE - Hospital de Santo António, Porto, Porto District
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, EPE, Vila Nova de Gaia, Porto District
  - Hospital Garcia de Orta, Almada, Setúbal District
  - Centro Hospitalar de Setúbal, Setúbal, Setúbal District
  - Hospital do Espírito Santo de Évora, EPE, Evora, Évora District

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bravo Baptista S, Pires de Morais G, Almeida Morais L, Costa J, Vinhas H, Campos G, Carrilho Ferreira P, Vale N, Seixo F, Santos M, Martins C, Rodrigues Bras D, Alexandre A, Raposo L. Anti-thrombotic and glucose lowering therapy in diabetic patients with coronary artery disease undergoing PCI with stent implantation: A prospective multicenter observational study on prescription patterns and clinical outcomes. Baseline inclusion data of the ARTHEMIS registry. Rev Port Cardiol. 2025 Sep;44(9):537-546. doi: 10.1016/j.repc.2025.03.006. Epub 2025 Jul 28. English, Portuguese. PMID 40738464